CLINICAL TRIAL: NCT05012800
Title: Safety and Immunogenicity of COVID-19 Vaccine Administered in Older Adults: A Multicenter Prospective Study
Brief Title: Safety and Immunogenicity of COVID-19 Vaccine Administered in Older Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: People's Hospital of Hunyuan County, Shanxi Province (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ky-2021-7-7-1
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Vaccine; Older Adults
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Vaccines in older adults (Experimental): Healthy people between the ages of 60 and 80 inoculated coronavirus vaccine on day 0 and day 21, respectively.
  Interventions: Biological: COVID-19 Vaccine
- COVID-19 Vaccines in young adults (Experimental): Healthy people between the ages of 20 and 59 inoculated coronavirus vaccine on day 0 and day 21, respectively.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Coronavirus vaccine was inoculated on day 0 and day 21, respectively.

SUMMARY:
The COVID-19 pandemic is causing unprecedented morbidity and mortality.The safe and effective Novel coronavirus vaccine is an effective means to block the transmission of the virus by building up the immune barrier of the population.Clinical studies have shown that elderly people are at high risk of severe COVID-19 infection and have poor clinical prognosis.Considering the current situation of aging population in China, the elderly people should be given priority to vaccinate to obtain protection and reduce the risk of novel coronavirus infection.However, the current data on vaccines are mostly from young and middle-aged healthy people, while there is little research data on COVID-19 vaccination in the elderly.This study mainly studied the safety and effectiveness of COVID-19 vaccine in the elderly population and explored its potential immune mechanism.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, controlled , open-label and phase I clinical trial. Older adults in the study included healthy people between the ages of 60 and 80 group. Those who is in line with the inclusion criteria and who is not in conformity with the exclusion criteria received two doses of COVID-19 vaccine at 0 days (baseline) and 21 days, respectively, and were followed up at 1, 3, 6, 9 and 12 months after completion of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* A COVID-19 vaccine is planned.
* Older adults subjects aged 60-80 years or young adults subjects aged 18-59 years.
* Able and willing to follow the requirements of the clinical trial protocol and complete the study follow-up for 12 months.
* HBsAg, anti-HCV, HIV and TPHA were negative.
* Body temperature ≤37.0℃.

Exclusion Criteria:

* People who are allergic to any component of the vaccine, or have a serious history of vaccine allergy.
* Women who is pregnant, breastfeeding, or planning to be pregnant within 6 months.
* Sufferring serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension can not be well controlled by drugs.
* Patients with severe chronic diseases or diseases can not be controlled well during the progress, such as asthma, diabetes, thyroid disease, etc.
* Patients with congenital or acquired angioedema / neuroedema.
* Patients with lymphoma, leukemia and other systemic malignancies.
* Patients with convulsions, epilepsy, encephalopathy, psychiatric disorders and other progressive neurological disorders, or a family history of them.
* Patients with acute attack of chronic diseases.
* During vaccination, immunomodulators, systemic cytotoxic drugs, immune checkpoint inhibitors (PD-1 / PDL-1 / CTLA-4, etc.) and cell therapy, including NK cells, cytokine induced killer cells, Dendritic cells, CTL and Stem cells infusion are required.
* Other conditions determined by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety of coronavirus vaccine | Within 2 months after the first dose of coronavirus vaccine
  Recorded the adverse effects after COVID-19 vaccination
Immunogenicity of coronavirus vaccine | Within 2 months after the first dose of coronavirus vaccine
  Detected the dynamics and titers of anti-SARS-CoV-2 antibodies

SECONDARY OUTCOMES:
Safety of coronavirus vaccine | Through study completion, an average of 13 months
  Recorded the adverse effects after COVID-19 vaccination
Immunogenicity | Through study completion, an average of 13 months
  Detected the dynamics and titers of anti-SARS-CoV-2 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes